CLINICAL TRIAL: NCT05493709
Title: An Open-label, Single Arm, Multicenter, Phase III Study on the Efficacy, Safety, and Pharmacokinetics of FP-001 42 mg Controlled Release in Patients With Central (Gonadotropin-Dependent) Precocious Puberty (Casppian Study)
Brief Title: Efficacy, Safety, and Pharmacokinetics of Leuprolide Mesylate in Subjects With Central Precocious Puberty
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: QPS Holdings LLC (Industry); Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP-001-CP-001
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Puberty; Precocious, Central
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FP-001 42 mg (Experimental): All subjects will be pediatric patients with central precocious puberty. They will be injected twice with a depot formulation containing 42 mg of Leuprolide. The first dose on day 0 the second dose on week 24 (six months apart).
  Interventions: Drug: Leuprolide Mesylate, Subcutaneous injection of 42 mg Leuprolide

INTERVENTIONS:
Drug: Leuprolide Mesylate, Subcutaneous injection of 42 mg Leuprolide — All subjects will be pediatric patients with central precocious puberty. They will be injected twice with a depot formulation containing 42 mg of Leuprolide. The first dose on day 0 the second dose on week 24 (six months apart).

SUMMARY:
The study will evaluate if Leuprolide Mesylate is safe and effective in the treatment of subjects with central (gonadotropin-dependent) precocious puberty, when administered as two injections six months apart.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single-arm study. All subjects will be pediatric patients with central precocious puberty judged to be candidates for GnRH (gonadotropin releasing hormone) analog therapy, and all will receive two injections of FP-001 42 mg six-month apart in an unblinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 2 to 8 years (inclusive) or males aged 2 to 9 years (inclusive).
2. Confirmed diagnosis of CPP within 12 months of Baseline Visit (Day 0) but have not received prior GnRHa treatment for CPP.
3. Pubertal-type LH response at 60 minutes post GnRHa stimulation test before treatment initiation > 5 mIU/mL.
4. Clinical evidence of puberty, defined as Tanner stage ≥ 2 for breast development in females or testicular volume ≥ 4 mL in males.
5. Willing and able to participate in the study.
6. Difference between bone age (Greulich and Pyle method) and chronological age ≥ 1 year.
7. Bone age < 13 years for girls and < 14 years for boys.
8. Signed Institutional Review Board/Independent Ethics Committee (IRB/IEC)-approved informed consent form (ICF) by one or both parents (per IRB/IEC requirements), by the custodial parent(s) or by the legal guardian(s) (if required).
9. Signed Assent by patients as per IRB/IEC requirements.

Exclusion Criteria:

1. Gonadotropin-independent (peripheral) precocious puberty: extra pituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroid secretion. This includes true CPP triggered by other conditions, such as congenital adrenal hyperplasia.
2. Prior or current GnRH treatment for CPP.
3. Non-progressing isolated premature thelarche.
4. Presence of an unstable intracranial tumor or an intracranial tumor requiring neurosurgery or cerebral irradiation. Patients with hamartomas or adenomas not requiring surgery are eligible.
5. Any other condition, chronic illness or treatment that, in the opinion of the Investigator, may interfere with growth or other study endpoints (e.g., chronic steroid use [except mild topical steroids], renal failure, diabetes, moderate to severe scoliosis, previously treated intracranial tumor).
6. Prior or current therapy with medroxyprogesterone acetate, growth hormone or insulin-like growth factor-1 (IGF-1).
7. Major medical or psychiatric illness that could interfere with study visits.
8. Diagnosis of short stature (i.e., 2.25 standard deviations (SD) below the mean height for age).
9. Positive urine pregnancy test.
10. Known hypersensitivity to GnRH or related compounds.
11. Any other medical condition or serious intercurrent illness that, in the opinion of the Investigator, may make it undesirable for the patients to participate in the study.
12. Any other condition(s) which could significantly interfere with Protocol compliance.
13. Treatment with an investigational product within 5 half-lives of that product in prior clinical studies before the baseline visit (Day 0).
14. Known history of seizures, epilepsy, and/or central nervous system disorders that may be associated with seizures or convulsions.
15. Prior (within 6 months of Baseline (Day 0)) or current use of medications that, per Investigator opinion, have been associated with seizures or convulsions.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Leuprolide Mesylate (FP-001 42 mg) | 48 weeks
  The percentage of patients with serum LH concentrations < 4 mIU/mL 60 minutes following an abbreviated GnRHa stimulation test at Visit 6 (Week 24).

SECONDARY OUTCOMES:
Effect of FP-001 42 mg on bone age progression | 24 and 48 weeks
  Evaluate the changes in bone age progression from the baseline to Weeks 24 and 48 using centralized analysis of wrist x-ray
Effect of FP-001 42 mg on growth rate | 48 weeks
  Evaluate the changes in growth rate and bone age advancement relative to chronological age from baseline to end of study using height in meters
Effect of FP-001 42 mg on physical signs of puberty | 48 weeks
  Evaluate the change in physical signs of puberty as measure by Tanner stages from baseline to end of study
Effect of FP-001 42 mg on suppression of physical signs of puberty | 48 weeks
  Evaluate the percentage of patients with suppression of physical signs of puberty
Acute-On-Chronic (AOC) phenomenon of serum testosterone and LH | 48 weeks
  Evaluate The proportion of subjects exhibiting "acute-on-chronic" phenomenon (i.e., related to the second dose of FP-001 42 mg)

CONTACTS AND LOCATIONS:
Overall Officials: Bassem Elmankabadi, Study Director — Foresee Pharma
Locations (41):
- United States (10):
  - Arizona University, Tucson, Arizona
  - Rady Children's Hospital- San Diego, San Diego, California
  - Nemours Children's Health Center, Jacksonville, Florida
  - Johns Hopkins - All Children's Hospital, St. Petersburg, Florida
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Indiana University, Indianapolis, Indiana
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's, Fort Worth, Texas
  - Virginia University, Charlottesville, Virginia
  - Multicare Health System, Tacoma, Washington
- China (24):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Children's Hospital affiliated to Capital Institute of Pediatrics, Beijing, Chaoyang District
  - The first Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Pearl River Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Wuhan Children's Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Children's Hospital of Shanxi, Taiyuan, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang
  - Ningbo Women & Children's Hospital, Ningbo, Zhejiang
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Children's Hospital of Fudan University, Shanghai
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
- University Pediatric Hospital, San Juan, Puerto Rico
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital-Kaohsiung branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - LinKou Chang-Gung Memorial Hospital (CGMH-LK), Taoyuan

IPD SHARING:
Plan to Share IPD: No